CLINICAL TRIAL: NCT07211633
Title: A Phase 3, Non-Inferiority, Randomized, Open-Label, Parallel Group, Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, Radiological and Clinical Effects of Subcutaneous Ublituximab Versus Intravenous Ublituximab in Patients With Multiple Sclerosis
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, Radiological and Clinical Effects of Subcutaneous Ublituximab in Participants With Relapsing Multiple Sclerosis (RMS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG1101-RMS-SC301; 2025-521127-73-00 (Other: EU CT Number)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ublituximab IV (Active Comparator): Approved dosage.
  Interventions: Biological: Ublituximab
- Ublituximab SC Regimen 1 (Experimental): New regimen.
  Interventions: Biological: Ublituximab
- Ublituximab SC Regimen 2 (Experimental): New regimen.
  Interventions: Biological: Ublituximab

INTERVENTIONS:
Biological: Ublituximab — Administered as an IV infusion.
  Other Names: TG-1101
  Arms: Ublituximab IV
Biological: Ublituximab — Administered as an SC injection.
  Other Names: TG-1101
  Arms: Ublituximab SC Regimen 1; Ublituximab SC Regimen 2

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of ublituximab when administered subcutaneously (SC) compared to intravenous (IV) administration in participants with RMS.

DETAILED DESCRIPTION:
This is a Phase 3, open label, parallel-group, multicenter study in participants with RMS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RMS (2017 Revised McDonald criteria).
2. Expanded Disability Status Scale (EDSS) score ≤ 5.5 at screening.
3. Neurologically stable for > 30 days prior to Screening and Day 1.
4. Female participants of childbearing potential must consent to use a highly effective method of contraception from consent and for 6 months after the last dose of ublituximab.

Exclusion Criteria:

1. Primary-progressive Multiple Sclerosis (PPMS) or inactive Secondary Progressive Multiple Sclerosis (SPMS).
2. Active chronic disease of the immune system other than MS or immunodeficiency syndrome.
3. Participants with significantly impaired bone marrow function or significant leukopenia or thrombocytopenia.
4. Participants who previously received anti-CD20 therapy at any time; any approved therapy to treat MS within 5 half-lives of the medication prior to screening.

Note: Other Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Week 0 to Week 24 (AUC0-W24) of Ublituximab | Up to Week 24

SECONDARY OUTCOMES:
Minimum Plasma Concentration (Cmin) of Ublituximab | Up to Week 24
Average Concentration at Steady State (Cavg,ss) of Ublituximab | Up to Week 120
Maximum Plasma Concentration (Cmax) of Ublituximab | Up to Week 120
Time to Maximum Plasma Concentration (Tmax) of Ublituximab | Up to Week 120
Last Observed Concentration (Clast) of Ublituximab | Up to Week 120
Area Under the Curve From Week 0 to Week 120 (AUC0-120) of Ublituximab | Up to Week 120
Concentration From Time 0 to Time of Last Concentration (AUClast) of Ublituximab | Up to Week 120
Time of Last Concentration (Tlast) of Ublituximab | Up to Week 120
Participants B Cell Counts | Up to Week 120
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to Week 120
Total Number of Gadolinium (Gd) enhancing T1 Lesions Per Magnetic Resonance Imaging (MRI) Scan | Up to Week 96
Total Number of New or Enlarging T2 lesions Per MRI Scan | Up to Week 96

CONTACTS AND LOCATIONS:
Locations (29):
- Bosnia and Herzegovina (4):
  - TG Therapeutics Investigational Trial Site, Banja Luka
  - TG Therapeutics Investigational Trial Site, Bihać
  - TG Therapeutics Investigational Trial Site, Mostar
  - TG Therapeutics Investigational Trial Site, Saravejo
- Bulgaria (4):
  - TG Therapeutics Investigational Trial Site, Pleven
  - TG Therapeutics Investigational Trial Site, Plovdiv
  - TG Therapeutics Investigational Trial Site, Sofia
  - TG Therapeutics Investigational Trial Site, Veliko Tarnovo
- Croatia (2):
  - TG Therapeutics Investigational Trial Site, Varaždin
  - TG Therapeutics Investigational Trial Site, Zagreb
- Czechia (6):
  - TG Therapeutics Investigational Trial Site, Brno
  - TG Therapeutics Investigational Trial Site, Hradec Králové
  - TG Therapeutics Investigational Trial Site, Jihlava
  - TG Therapeutics Investigational Trial Site, Ostrava
  - TG Therapeutics Investigational Trial Site, Pardubice
  - TG Therapeutics Investigational Trial Site, Zlín
- TG Therapeutics Investigational Trial Site, Tbilisi, Georgia
- Hungary (4):
  - TG Therapeutics Investigational Trial Site, Budapest
  - TG Therapeutics Investigational Trial Site, Kaposvár
  - TG Therapeutics Investigational Trial Site, Kistarsca
  - TG Therapeutics Investigational Trial Site, Pécs
- North Macedonia (2):
  - TG Therapeutics Investigational Trial Site, Shtip
  - TG Therapeutics Investigational Trial Site, Skopje
- Ukraine (6):
  - TG Therapeutics Investigational Trial Site, Cherkasy
  - TG Therapeutics Investigational Trial Site, Ivano-Frankivsk
  - TG Therapeutics Investigational Trial Site, Kyiv
  - TG Therapeutics Investigational Trial Site, Lviv
  - TG Therapeutics Investigational Trial Site, Ternopil
  - TG Therapeutics Investigational Trial Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: No